CLINICAL TRIAL: NCT04925778
Title: An Open-label, Observational Study in Patients With Relapsing-Remitting Multiple Sclerosis Switched to Bafiertam® (Monomethyl Fumarate) From Dimethyl Fumarate (PERSIST)
Brief Title: Observational Study in Patients With Relapsing-Remitting Multiple Sclerosis Switched to Bafiertam® From Dimethyl Fumarate
Acronym: PERSIST
Status: Withdrawn | Type: Observational
Why Stopped: Business considerations
Sponsor: Banner Life Sciences LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BLS-11-403
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Bafiertam; Tecfidera; dimethyl fumarate; monomethyl fumarate; gastrointestinal
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — monomethyl fumarate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: monomethyl fumarate — Patients will be prescribed 190 mg (two 95 mg capsules) self-administered twice/day,
  Other Names: Bafiertam®, BLS-11

SUMMARY:
This is an open-label, multicenter, observational study evaluating GI symptoms in relapsing-remitting multiple sclerosis (RRMS) patients who switch from dimethyl fumarate (DMF) to Bafiertam®.

DETAILED DESCRIPTION:
This is an open-label, multicenter, observational study evaluating GI symptoms in relapsing-remitting multiple sclerosis (RRMS) patients who switch from dimethyl fumarate (DMF) to Bafiertam® (monomethyl fumarate).

Adult patients with a diagnosis of RRMS receiving continuous treatment with DMF monotherapy and who are experiencing GI symptoms will be eligible to enroll in the study.

Patients will be identified and screened by chart review and invited to report GI Symptoms for one baseline week using a study app downloaded on their own smartphone/tablet. During this week, patients will continue their currently prescribed and remaining DMF treatment and will record their GI symptoms daily using the app.

At the end of the Baseline Period, patients will be asked to cease administration of the DMF, and to commence self-treatment with Bafiertam® 95 mg capsules twice a day (total daily dose of 380 mg) approximately 12 hours apart the following day for 28 days. They will be required to continue to record their GI symptoms each day.

On Day 28; End-of Study [EOS]) the patient's diary will be reviewed, adverse events (AE) recorded, and drug accountability performed.

Following EOS patients will be asked if they wish to continue Bafiertam® treatment. Those patients who elect to continue will be contacted one month and two months after EOS to ascertain if they remain on Bafiertam®.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or non-pregnant female aged 18years and older.
2. Diagnosis of RRMS (per McDonald 2010 Criteria) at screening [Polman 2011].
3. Currently being treated with dimethyl fumarate (DMF; Tecfidera® or generic equivalent). At least 1 week and 1 day of continuous treatment with DMF monotherapy prior to initiation of Bafiertam®. Note: continuous treatment with DMF is defined as treatment uninterrupted by other disease-modifying treatment.
4. GI symptoms (defined as any combination of abdominal pain, nausea, vomiting, diarrhea, constipation, bloating, or flatulence) while receiving treatment with DMF.
5. Must be naïve to Bafiertam®.
6. Additional inclusion criteria apply

Key Exclusion Criteria:

1. Diagnosis of primary progressive, secondary progressive, or progressive relapsing MS (as defined by Lublin and Reingold) [Lublin 2014].
2. Females breastfeeding, pregnant, or planning to become pregnant; or women who have a positive pregnancy test result during screening.
3. History of severe hypersensitivity (e.g., anaphylaxis or anaphylactoid reactions) to the active ingredient (monomethyl fumarate), dimethyl fumarate, diroximel fumarate (Vumerity®), or any of the excipients.
4. Lymphocyte counts less than 1000/microliter. Any other clinically significant abnormalities in CBC, blood and urine chemistries, or liver function tests in the past 30 days.
5. History of severe opportunistic infections (including progressive multifocal leukoencephalopathy (PML) and herpes zoster) or any clinically significant, cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic (other than MS), dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator.
6. Any prior suspicion of PML.

9. Additional exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of relapsing-remitting multiple sclerosis currently treated with dimethyl fumarate (DMF), and experiencing gastrointestinal symptoms attributable to DMF are eligible. Sufficient patients will be enrolled until 50 evaluable patients complete the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-29 (Estimated)

PRIMARY OUTCOMES:
Comparison of the frequency and severity of GI symptoms before and after switching to Bafiertam®. | 28 days
  The GI tolerability of Bafiertam® following a switch from dimethyl fumarate will be assessed by determining the frequency and severity of GI events using a modified gastrointestinal symptom scale.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Lategan, D.Phil., Study Director — Banner Life Sciences LLC

IPD SHARING:
Plan to Share IPD: No